CLINICAL TRIAL: NCT05021510
Title: Effects of Simultaneous Traction and Neural Mobilization on Pain and Function in Cervical Radiculopathy.
Brief Title: Simultaneous Traction and Neural Mobilization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/01030 Sabah
Record Dates: First submitted 2021-08-23; First posted 2021-08-25 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Cervical Radiculopathy
MeSH Terms: conditions — Radiculopathy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Simultaneous Cervical Traction & Neural Mobilization (Experimental): Traction is a maneuver of distracting force to the cervical spine to cervical segments/grants decompression of nerve roots. For traction, 10% of the total body weight would be taken. Previous researches that investigated cervical traction found adequate effectiveness on pain reduction in neck and arm as well as improvement in nerve function parameters, and enhancement in neck mobility. The patient would be placed in a supine lying position with the cervical spine placed at 15º of flexion. The head strap will be fitted under the patient's occiput and chin. A safety switch will be given to the patient and ask him to press it if he would feel any kind of discomfort.
  Interventions: Other: Simultaneous Cervical Traction & Neural Mobilization
- consecutive Cervical Traction & Neural Mobilization (Active Comparator): the same description is for active comparator except for treatment mode to consecutive.
  Interventions: Other: consecutive Cervical Traction & Neural Mobilization

INTERVENTIONS:
Other: Simultaneous Cervical Traction & Neural Mobilization — Simultaneously Mechanical Cervical traction with Neural Mobilization of the upper limb for 3 times a week, 45 minutes per day for 4 weeks
  Arms: Simultaneous Cervical Traction & Neural Mobilization
Other: consecutive Cervical Traction & Neural Mobilization — consecutive Mechanical Cervical traction with Neural Mobilization of the upper limb for 3 times a week, 45 minutes per day for 4 weeks
  Arms: consecutive Cervical Traction & Neural Mobilization

SUMMARY:
Neck pain is a frequently reported complaint of the musculoskeletal system which generally has a huge impact on health care expenditure; ascribed to visits to health care providers, disability, and sick leaves. A variety of manual therapy techniques including Cervical traction (CT) and neural mobilization techniques (NMTs) have been prescribed in the management of CR because of their immediate analgesic effect. Both techniques have been proposed to reduce pain and functional limitations in CR. Traction increases the separation of the vertebral bodies which eventually reduces the central pressure in the disk space and encourages the disk nucleus to get back to a central position. The current literature lends assistance to the utilization of the traction in addition to other physical therapy procedures for pain reduction, with less significant impact on function and disability. Further studies should investigate to explore the most effective traction method and dosage, the subgroups of patients with CR, or the pain stage (acute, subacute, or chronic) most benefited by this intervention and the physical therapy procedures that yield the most effective outcomes when combined with traction.

DETAILED DESCRIPTION:
Researchers have started exploring that neural tissue mobilization along with conventional treatment is more effective in decreasing pain and improving cervical range of motion and mental component of quality of life in unilateral cervical radiculopathy (CR) patients than intermittent cervical traction and conventional treatment. Future randomized controlled trials are warranted with the purpose to compare the long-term effectiveness of cervical traction with neural mobilization in CR, as well as the effect of these two techniques in comparison with other interventions. Some literature recommended the simultaneous application of mechanical cervical traction along with neural mobilization in the treatment of Unilateral Cervical Radiculopathy. There are numerous studies in which both groups received Cervical traction (CT) and neural mobilization (NM) was added in only one group along with cervical traction or studies in which both groups received NM and CT was administered in only one group as well, there are also some studies in which one group received only CT and other group received only NM but there isn't any study yet in which we can compare the effect of simultaneous administration of CT and NM and consecutive administration of CT and NM.

Pain and functional limitation in cervical radiculopathy can be treated with mechanical cervical traction and neural mobilization. The purpose of the study is to determine that is simultaneous administration of cervical traction and neural mobilization is more effective than consecutive administration in the management of cervical radiculopathy. The findings of the study will provide an insight into the low-cost evidence-based conservative management of cervical radiculopathy.

ELIGIBILITY:
Inclusion Criteria:

* Participants with Chronic Cervical Radiculopathy for 6 months will be included.
* Participants with Positive Spurling and Upper Limb Neural Tension Tests (ULNTTs) will be included.
* Participants of age 20 to 60 will be included

Exclusion Criteria:

* The participants with cervical myelopathy and other pathologies will not be included.
* The participants with Vertigo/dizziness will not be included.
* The participants with bilateral symptoms will not be included.
* The participants with other musculoskeletal conditions in the affected limb will not be included.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-08-15 (Actual); Primary Completion 2022-08-20 (Actual); Study Completion 2022-08-20 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | week 4
  NPRS for pain is a unidimensional measure of pain intensity. Similar to visual analogue scale (VAS), the NPRS is anchored by describing pain severity extremes. The NPRS can be administered verbally or graphically for self-completion.
Neck Disability Index (NDI) for function | week 4
  NDI used to measure cervical pain and functional disability. The NDI was created using a questionnaire with 10 questions based on the Oswestry Index, which evaluates restrictions to ordinary life in relation to lumbar pain. The subjects selected a score of one to six (0 to 5) in 10 items: reading, headache, concentration, work, driving, sleeping, leisure life, pain intensity, ordinary life, and raising an object.
  The higher the sum of each item's score, the more severe the functional disability related to cervical abnormality. Zero to four points, five to 14 points, 15 to 24 points, 25 to 34 points, and 35 points or higher signify no disability, weak disability, moderate disability, severe disability, and complete disability, respectively
Short Form Quality of Life 12: (physical, mental) | week 4
  The developers of short form (SF) 36 have consequently, suggested that a 12 item sub-set of the items may accurately reproduce the two summary component scores which can be derived from the SF 36 [the physical component score (PCS) and the mental component score (MCS)].
  The scores were put in the free online orthopedic calculator "ortho tool kit" and two summary scores have been generated: Physical component score and mental component score.

CONTACTS AND LOCATIONS:
Overall Officials: Arshad Malik, PhD, Principal Investigator — Riphah International University
Locations (1):
- The Physiotherapy Clinic, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cohen SP. Epidemiology, diagnosis, and treatment of neck pain. Mayo Clin Proc. 2015 Feb;90(2):284-99. doi: 10.1016/j.mayocp.2014.09.008. PMID 25659245
- [Background] Ayub A, Osama M, Ahmad S. Effects of active versus passive upper extremity neural mobilization combined with mechanical traction and joint mobilization in females with cervical radiculopathy: A randomized controlled trial. J Back Musculoskelet Rehabil. 2019;32(5):725-730. doi: 10.3233/BMR-170887. PMID 30664500
- [Background] Savva C, Korakakis V, Efstathiou M, Karagiannis C. Cervical traction combined with neural mobilization for patients with cervical radiculopathy: A randomized controlled trial. J Bodyw Mov Ther. 2021 Apr;26:279-289. doi: 10.1016/j.jbmt.2020.08.019. Epub 2020 Sep 2. PMID 33992259
- [Background] Tarazona D, Boody B, Hilibrand AS, Stull J, Bell K, Fang T, Goyal D, Galetta M, Kaye D, Kepler CK, Kurd MF, Woods BI, Radcliff KE, Rihn JA, Anderson DG, Vaccaro AR, Schroeder GD. Longer Preoperative Duration of Symptoms Negatively Affects Health-related Quality of Life After Surgery for Cervical Radiculopathy. Spine (Phila Pa 1976). 2019 May 15;44(10):685-690. doi: 10.1097/BRS.0000000000002924. PMID 30395087
- [Background] Efstathiou MA, Stefanakis M, Savva C, Giakas G. Effectiveness of neural mobilization in patients with spinal radiculopathy: a critical review. J Bodyw Mov Ther. 2015 Apr;19(2):205-12. doi: 10.1016/j.jbmt.2014.08.006. Epub 2014 Aug 17. PMID 25892373
- [Background] Romeo A, Vanti C, Boldrini V, Ruggeri M, Guccione AA, Pillastrini P, Bertozzi L. Cervical Radiculopathy: Effectiveness of Adding Traction to Physical Therapy-A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Phys Ther. 2018 Apr 1;98(4):231-242. doi: 10.1093/physth/pzy001. PMID 29315428
- [Background] Caridi JM, Pumberger M, Hughes AP. Cervical radiculopathy: a review. HSS J. 2011 Oct;7(3):265-72. doi: 10.1007/s11420-011-9218-z. Epub 2011 Sep 9. PMID 23024624